CLINICAL TRIAL: NCT00926523
Title: Biomarkers in the Evaluation of Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Arunabh Talwar M.D., North Shore LIJ Health System
Other Study IDs: GCRC 0274
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Interstitial Lung Disease
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Interstitial Lung Disease; MIF
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Lung Diseases, Interstitial | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breathe condensate.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Controls: Subjects are made up of healthy adults
  Interventions: Other: Blood Gas; Other: Pulmonary Exercise Test; Other: Spirometry; Other: Breath Condensate Collector
- Affected: Subjects have Pulmonary Hypertension
  Interventions: Other: Blood Gas; Other: Pulmonary Exercise Test; Other: Spirometry; Other: Breath Condensate Collector

INTERVENTIONS:
Other: Blood Gas — Subject will have both venous and arterial blood draws to assess for the bloods content of MIF
Other: Pulmonary Exercise Test — Subject will ride exercise bike to assess their pulmonary function level.
Other: Spirometry — To assess subjects lung function
Other: Breath Condensate Collector — Subject with use breathing apparatus to allow researchers to collect breath condensate to assess level of MIF in breathe condensate.

SUMMARY:
We hypothesize that hypoxia-induced pulmonary vascular remodeling is mediated by macrophage migration inhibitory factor (MIF), that remodeling is in fact the reflection of a chronic inflammatory process, and that MIF may be a useful biomarker of the severity and progression of both ILD and PH.

DETAILED DESCRIPTION:
We hypothesize that hypoxia-induced pulmonary vascular remodeling is mediated by macrophage migration inhibitory factor (MIF), that remodeling is in fact the reflection of a chronic inflammatory process, and that MIF may be a useful biomarker of the severity and progression of both ILD and PH.

To study this hypothesis, we have two specific aims:

1. To evaluate plasma MIF concentration as a marker of severity in ILD and PH and
2. To determine the utility of breathe condensate analysis in the evaluation of ILD and PH. If we are successful in identifying MIF as a biomarker, it may identify MIF as a useful therapeutic target, as we have shown in other inflammatory disorders.

ELIGIBILITY:
Inclusion Criteria:

* Subject are at least 18 years of age
* Subject has confirmed Pulmonary Hypertension and Interstitial Lung Disease
* Subject are able to complete study procedures, such as spirometry, and Pulmonary Exercise test.

Exclusion Criteria:

* Subject are pregnant
* Subject is unable to perform tasks associated with study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are either a healthy volunteer, or someone who has confirmed Pulmonary Hypertension and Interstitial Lung Disease
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arunabh Talwar, M.D., Principal Investigator — Northwell Health; Ed Miller, Ph.D, Principal Investigator — North Shore Long Island Jewish Healthy System
Locations (1):
- Interstitial Lung Disease and Pulmonary Hypertension Programs, New Hyde Park, New York, United States